CLINICAL TRIAL: NCT07190833
Title: A Phase 1 Study of OTS-412 (Recombinant Oncolytic Vaccinia Virus) in Combination With Hydroxyurea or Hydroxyurea/Atezolizumab in Treatment-refractory Solid Tumor Patients
Brief Title: A Phase 1 Study of OTS-412 (Recombinant Oncolytic Vaccinia Virus) in Treatment-refractory Solid Tumor Patients (South Korea)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bionoxx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OTS412-101(ROK)
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Treatment-Refractory Solid Tumors
MeSH Terms: interventions — Hydroxyurea; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): OTS412 1 * 10E8 pfu
  Interventions: Drug: OTS-412
- Cohort 2 (Experimental): OTS412 1 * 10E8 pfu + HU 15mg/kg/day
  Interventions: Drug: OTS-412; Drug: Hydroxyurea (HU)
- Cohort 3 (Experimental): OTS412 1 * 10E8 pfu + HU 25mg/kg/day
  Interventions: Drug: OTS-412; Drug: Hydroxyurea (HU)
- Cohort 4 (Experimental): OTS412 1 * 10E8 pfu + HU 35mg/kg/day
  Interventions: Drug: OTS-412; Drug: Hydroxyurea (HU)
- Cohort 5 (Experimental): OTS412 1 * 10E8 pfu + HU optimal dose + Atezolizumab 1200mg
  Interventions: Drug: OTS-412; Drug: Hydroxyurea (HU); Drug: Atezolizumab
- Cohort 6 (Experimental): OTS412 3 * 10E8 pfu + HU optimal dose + Atezolizumab 1200mg
  Interventions: Drug: Hydroxyurea (HU); Drug: Atezolizumab; Drug: OTS-412
- Expansion cohort (Experimental): OTS412 optimal dose + HU optimal dose + Atezolizumab 1200mg
  Interventions: Drug: Hydroxyurea (HU); Drug: Atezolizumab; Drug: OTS-412

INTERVENTIONS:
Drug: OTS-412 — 1×10E8 pfu, once, 1 cycle, IT
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: Hydroxyurea (HU) — 15 mg/kg/day, 14 days, 1 cycle, PO
  Arms: Cohort 2
Drug: Hydroxyurea (HU) — 25 mg/kg/day, 14 days, 1 cycle, PO
  Arms: Cohort 3
Drug: Hydroxyurea (HU) — 35 mg/kg/day, 14 days, 1 cycle, PO
  Arms: Cohort 4
Drug: Hydroxyurea (HU) — optimal dose, 14 days, 1 cycle, PO
  Arms: Cohort 5; Cohort 6; Expansion cohort
Drug: Atezolizumab — 1,200 mg, once, 1 cycle, IV
  Arms: Cohort 5; Cohort 6; Expansion cohort
Drug: OTS-412 — 3×10E8 pfu, once, 1 cycle, IT
  Arms: Cohort 6
Drug: OTS-412 — optimal dose, once, 1 cycle, IT
  Arms: Expansion cohort

SUMMARY:
This clinical trial aims to determine whether the administration of the investigational drug OTS-412, OTS-412 in combination with hydroxyurea or hydroxyurea/atezolizumab is safe and effective for patients with various types of cancer.

DETAILED DESCRIPTION:
The primary objective of this study is:

* to evaluate the safety of OTS-412 monotherapy, combination therapy of OTS-412 and hydroxyurea, or combination therapy of OTS-412, hydroxyurea, and atezolizumab
* to find an optimal dosage of hydroxyurea when used in combination with OTS 412. Hydroxyurea is currently used at dosages of 15-35 mg/kg/day for certain conditions, and the optimal dosage when combined with the oncolytic virus will be determined within this range.
* to find an optimal dosage of OTS-412 when used in combined with hydroxyurea and atezolizumab.

The secondary objectives include evaluating anti-tumor effects, immune responses, and pharmacokinetics (PK) of OTS-412 in blood over time after administration.

This study focuses on various solid tumors that are resistant to standard therapies, particularly immune checkpoint inhibitors alone or in combination with other therapies.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. Diagnosed with a malignant solid tumor via histology or cytology, although a radiological diagnosis is permissible for hepatocellular carcinoma
3. Solid tumors that demonstrate limited response or resistant to SOC therapy, particularly when atezolizumab or other PD-L1 inhibitors, or PD-1 inhibitors are administered as monotherapy or in combination therapy. This may include, but not limited to, hepatocellular carcinoma, melanoma, renal cell carcinoma, urothelial carcinoma, biliary cancer, head and neck cancer, gastric cancer, breast cancer, colorectal cancer, and any solid tumor with microsatellite instability (MSI)-high status. At minimum, SOC treatment presented in the Protocol should have been received for each cancer type.
4. Patients with tumors that have known actionable molecular alterations (i.e. EGFR, ALK, BRAF, etc) must have progressed on targeted therapy.
5. Lesions that are deemed feasible for injection either directly (palpable subcutaneous tumors) or under ultrasound guidance (deep-seated tumors). Additionally, tumor(s) should not be adjacent or encasing vital structures such as major nerves or blood vessels, pericardium, gastrointestinal tract or other hollow organs, mucosal regions or spinal cord that could cause occlusion or compression in case of tumor swelling or erosion and major bleeding in the case of necrosis.
6. At least one measurable (longest diameter, LD ≥1 cm) and injectable tumor that has not been previously received local treatment on computed tomography (CT) or magnetic resonance imaging (MRI)
7. The total volume of injectable tumor(s) should be 2 cm3 or more in 1x10E8 pfu dosing cohorts and 6 cm3 or more in 3x10E8 pfu dosing cohorts.
8. Life expectancy of 12 weeks or more
9. Eastern cooperative oncology group (ECOG) performance status is 0, 1, or 2
10. Adequate pulmonary function, such as baseline pulse oximetry of at least 92% on room air
11. Laboratory test results meet the following:

    * ANC ≥ 1,500 /μL
    * White blood cell (WBC) ≥ 2,500 /μL
    * Hemoglobin (Hb) ≥ 9.0 g/dL without packed red blood cell transfusion within the prior 2 weeks
    * Platelet ≥ 75,000 /μL without platelet transfusion
    * AST and ALT ≤ 5 × ULN
    * Total bilirubin ≤ 1.5 × ULN
    * Creatinine clearance ≥ 60 mL/minute (measured using Cockcroft-Gault formula).
    * LDH ≤ 3 × ULN
    * INR or aPTT ≤ 1.5 × ULN.
12. Voluntarily decided to participate in this clinical study and provided written consent

Exclusion Criteria:

1. Patients who have previously received talimogene laherparepvec (Imlygic) or any other oncolytic virus, have received any systemic or local anti-cancer therapy for tumors within 4 weeks prior to the first administration of the study drugs(C1D1), or have not recovered from the adverse events due to these therapies to at least Grade 1 severity or returned to baseline levels prior to C1D1, with the exceptions of any grade of alopecia and Grade 2 neuropathy.
2. Patients who have untreated symptomatic brain metastases, have treated brain metastases without evidence of stability or improvement on two scans at least two weeks apart, have leptomeningeal disease regardless of treatment, or have received anti-convulsants within the last 28 days.
3. Tumors adjacent to vital neurovascular structures or at risk of airway compromise in the event of post injection tumor swelling, bleeding, or inflammation. Patients with tumors near vital structures can be enrolled as long as they have other lesions that are appropriate for injection (these tumors near vital structures will not be injected).
4. History of other malignancies that developed within 5 years (However, cervical carcinoma in situ, basal cell carcinoma, or squamous cell skin cancer, and all cancers after 5 years since it was cured are acceptable.)
5. History of organ transplant surgery
6. Known significant immunodeficiency due to underlying illness (e.g., HIV/AIDS) and/or immune-suppressive medication including high-dose systemic corticosteroids (prednisone 20 mg/day or equivalent which is ongoing and/or was taken more than 4 weeks within the preceding 2 months of study treatment)
7. History of or active autoimmune disease
8. Ongoing severe inflammatory skin disease (as determined by the Investigator) requiring medical treatment or history of severe eczema (as determined by the Investigator) requiring prior medical treatment
9. Anticoagulation or anti-platelet medication that cannot be withheld for the required period prior to and after the OTS-412 injection, specifically:

   * Coumadin for 7 days
   * Direct Factor Xa inhibitor (rivaroxaban, apixaban, edoxaban) for 4 days
   * Oral direct thrombin inhibitor (dabigatran) for 4 days
   * Aspirin, clopidogrel, ticagrelor for 7 days
   * Prasugrel for 9 days
   * Low molecular weight heparin for 24 hours
   * Unfractionated heparin for 12 hours Please contact the Sponsor for questions regarding the management of other antithrombotic agents prior to treatment.
10. Taking antiviral drugs (immunoglobulin, interferon, etc.) or being unable to discontinue these medications at least 7 days prior to receiving the study drugs (note that oral antiviral drugs for hepatitis B and C are allowed).
11. Severe medical conditions, as determined by the Investigator, that may increase the patient's susceptibility to adverse medical risks during or after OTS-412 treatment, such as volume loading, tachycardia, or hypotension.
12. Current or history of significant cardiovascular disease, including significant coronary artery disease (e.g., requiring angioplasty or stent), congestive heart failure within the preceding 12 months, myocardial infarction, ischemic cardiomyopathy, or myocarditis, unless cardiology consultation and clearance have been obtained for study participation
13. History of the side effects of past smallpox vaccinations
14. History of the hypersensitivity or severe/serious AEs to the components of the study drugs
15. Unable to receiving a contrast medium for a radiological scan due to a history of allergy to iodide contrast agents
16. Vaccination with live vaccines within 4 weeks before the first administration of the study drugs
17. Receiving an investigational product within 4 weeks prior to the first administration of the study drugs
18. Pregnant or breastfeeding women
19. Patient who does not consent to the use of appropriate contraceptive methods for at least 6 months, when the woman is of childbearing age, or at least 1 year, when the male patient's spouse is a woman of childbearing age, after the last administration of the study drugs
20. Other medical condition that in the judgement of the Investigator may increase the risk associated with study participation or may interfere with interpretation of study results and/or otherwise make the patient inappropriate for study participation
21. Patient unable or unwilling to comply with the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 or higher in OTS 412, OTS-412/HU combination, and OTS 412/HU/atezolizumab combination treatment | From enrollment to 180 days after the last dose of the study drugs.

SECONDARY OUTCOMES:
Tumor response, as determined by the Investigator according to RECIST v1.1 (or mRECIST for hepatocellular carcinoma) and/or iRECIST | From enrollment to 28 days after the last dose of the study drugs
Overall survival defined as time from the study drug initiation to death from any cause | From enrollment up to 15 years after end of study
PK analysis: Assessment of the concentration of OTS-412 genomic particles (qPCR) in blood over time | From enrollment to Day 22
Rate of patients to achieve target absolute neutrophil count (ANC) level (between 1500 and 3000/μL) 7 days after OTS-412 administration | 7 days after OTS-412 administration
Changes in ANC over time | From enrollment to 180 days after the last dose of the study drugs.
Changes in lymphocytes count over time | From enrollment to 180 days after the last dose of the study drugs.
Changes in immunophenotype of lymphocytes over time | From enrollment to Day 22
Changes in serum cytokines (including but not limited to IL-1β, IL-6, INF-γ, TNF-α) over time | From enrollment to Day 22
Assessment of tumor tissue histology and immunology, including immunological assays for T cells and programmed cell death ligand 1 (PD-L1) expression (optional) | From enrollment to Day 22(exceptionally, for Cohort 1, 28 days after last study drug administration)
Viral shedding analysis: Assessment of the presence of the virus in oral and urine samples | From enrollment to Day 22
Neutralizing antibody measurement against OTS-412 | From enrollment to Day 22
Firefly luciferase (FLuc) T cell response assessment | From enrollment to Day 22

OTHER OUTCOMES:
Changes in activated neutrophils (aN) and activated T lymphocytes (aT) assessed by FLuc activity in isolated neutrophils and T lymphocytes over time | From enrollment to Day 22